CLINICAL TRIAL: NCT02962713
Title: Giomer vs Glass Ionomer Cement for ART Occlusoproximal Restorations: a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniela Prócida Raggio, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GIOMERART
Record Dates: First submitted 2016-08-30; First posted 2016-11-11 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries
Keywords: Atraumatic Restorative Treatment; glass ionomer cement; primary teeth; dental caries.
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ART with Equia (Active Comparator): Occlusal-proximal restoration in primary molars using Equia (Easy/Quick/Unique/Intelligent/Aesthetic) from GC Corp, encapsulated, pre-dosed and mechanized handling.
  Interventions: Procedure: ART with Equia
- ART with Giomer Beautifil-Bulk Restorative (Experimental): Occlusal-proximal restoration in primary molars using Giomer Beautifil-Bulk Restorative (SHOFU Inc)
  Interventions: Procedure: ART with Giomer Beautifil-Bulk Restorative

INTERVENTIONS:
Procedure: ART with Equia — Occlusal-proximal ART restorations in primary molars using Equia (Easy/Quick/Unique/ Intelligent/Aesthetic) will be performed. No local anesthesia will be used. Infected carious tissue will be removed with hand instruments, and the cavities restored with GIC (Glass Ionomer Cement). The cavity will be filled with GIC. After the press-finger technique, the excess of material will be removed and occlusion will be checked.
  Arms: ART with Equia
Procedure: ART with Giomer Beautifil-Bulk Restorative — Occlusal-proximal ART restorations in primary molars using Giomer will be performed. No local anesthesia will be used. Infected carious tissue will be removed with hand instruments, and the cavities restored with Giomer Beautifil-Bulk Restorative and occlusion will be checked.
  Arms: ART with Giomer Beautifil-Bulk Restorative

SUMMARY:
Although the Atraumatic Restorative Treatment (ART) is well settled in the literature regarding occlusal-proximal cavities, the longevity of these restorations is still lower when compared to occlusal ones. This factor is often associated with low mechanical properties of glass ionomer cements (GIC). The objective of this randomized clinical trial is to evaluate the long-term cost-effectiveness of two different materials: an encapsulated GIC - Equia (GC Corp), compared with Giomer (Beautifill Bulk Restorative - Shofu) used as restoratives materials in occlusal-proximal ART restorations of primary molars. Children aged between 4 and 8 years, will be selected in schools in the city of Cerquilho, São Paulo. All restorations will be held following the precepts of the ART and the manufacturer's instructions. The restorations will be evaluated after 3, 6, 12, 18 and 24 months according to Roeleveld et al. (2006) criteria. To verify the survival of the restorations will be used Kaplan-Meier survival analysis and log rank test. To evaluate the association between the clinical variables, Cox regression test will be applied. For the cost analysis will be used analysis of variance. The level of significance for all tests will be considered to 5%.

ELIGIBILITY:
Inclusion Criteria:

* Children aging between 4 and 8 years
* Children presenting good health conditions
* Children whose parents or legal guardians accept and sign the consent form
* Children with at least one occlusal proximal caries lesion in primary molars
* only occlusal-proximal surfaces with caries lesions with dentin involvement

Exclusion Criteria:

* severe behavioral issues
* presence of fistula or abscess near the selected tooth
* presence of pulp exposure in the selected tooth
* presence of mobility in the selected tooth

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Longevity of atraumatic restoration using Roeleveld et al. (2006) criteria | up to 24 months
  The treatments will be classified as successful when they present a clinical satisfactory aspect. Otherwise, "minor failure" will be analyzed. "Minor failures" are those in which there is a defect in the restoration, but it does not interfere in the tooth health.

SECONDARY OUTCOMES:
Cost-effiectiveness assessment | an average of 24 months
  The direct cost analysis of the ART performed with the encapsulated GICs will be based on previous publications (Takanashi et al., 2004; Oscarson et al., 2003) adjusted to the Brazilian reality (Floriano et al., 2013). For this, we will consider professional cost and cost of the procedure itself.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Raggio, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walsh T, Worthington HV, Glenny AM, Appelbe P, Marinho VC, Shi X. Fluoride toothpastes of different concentrations for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD007868. doi: 10.1002/14651858.CD007868.pub2. PMID 20091655
- [Background] van 't Hof MA, Frencken JE, van Palenstein Helderman WH, Holmgren CJ. The atraumatic restorative treatment (ART) approach for managing dental caries: a meta-analysis. Int Dent J. 2006 Dec;56(6):345-51. doi: 10.1111/j.1875-595x.2006.tb00339.x. PMID 17243467
- [Background] ten Berge M, Hoogstraten J, Veerkamp JS, Prins PJ. The Dental Subscale of the Children's Fear Survey Schedule: a factor analytic study in The Netherlands. Community Dent Oral Epidemiol. 1998 Oct;26(5):340-3. doi: 10.1111/j.1600-0528.1998.tb01970.x. PMID 9792126
- [Background] Takanashi Y, Penrod JR, Lund JP, Feine JS. A cost comparison of mandibular two-implant overdenture and conventional denture treatment. Int J Prosthodont. 2004 Mar-Apr;17(2):181-6. PMID 15119869
- [Background] Sunico MC, Shinkai K, Katoh Y. Two-year clinical performance of occlusal and cervical giomer restorations. Oper Dent. 2005 May-Jun;30(3):282-9. PMID 15986946
- [Background] Shimazu K, Oguchi R, Takahashi Y, Konishi K, Karibe H. Effects of surface reaction-type pre-reacted glass ionomer on oral biofilm formation of Streptococcus gordonii. Odontology. 2016 Sep;104(3):310-7. doi: 10.1007/s10266-015-0217-2. Epub 2015 Aug 30. PMID 26319990
- [Background] Sheiham A. Dental caries affects body weight, growth and quality of life in pre-school children. Br Dent J. 2006 Nov 25;201(10):625-6. doi: 10.1038/sj.bdj.4814259. PMID 17128231
- [Background] Sengul F, Gurbuz T. Clinical Evaluation of Restorative Materials in Primary Teeth Class II Lesions. J Clin Pediatr Dent. 2015 Summer;39(4):315-21. doi: 10.17796/1053-4628-39.4.315. PMID 26161601
- [Background] Schriks MC, van Amerongen WE. Atraumatic perspectives of ART: psychological and physiological aspects of treatment with and without rotary instruments. Community Dent Oral Epidemiol. 2003 Feb;31(1):15-20. doi: 10.1034/j.1600-0528.2003.00021.x. PMID 12542428
- [Background] Santamaria R, Innes N. Trial shows partial caries removal is an effective technique in primary molars. Evid Based Dent. 2014 Sep;15(3):81-2. doi: 10.1038/sj.ebd.6401044. PMID 25343394
- [Background] Roeleveld AC, van Amerongen WE, Mandari GJ. Influence of residual caries and cervical gaps on the survival rate of Class II glass ionomer restorations. Eur Arch Paediatr Dent. 2006 Jun;7(2):85-91. doi: 10.1007/BF03320820. PMID 17140533
- [Background] Raggio DP, Hesse D, Lenzi TL, Guglielmi CA, Braga MM. Is Atraumatic restorative treatment an option for restoring occlusoproximal caries lesions in primary teeth? A systematic review and meta-analysis. Int J Paediatr Dent. 2013 Nov;23(6):435-43. doi: 10.1111/ipd.12013. Epub 2012 Nov 28. PMID 23190278
- [Background] Phantumvanit P, Songpaisan Y, Pilot T, Frencken JE. Atraumatic restorative treatment (ART): a three-year community field trial in Thailand--survival of one-surface restorations in the permanent dentition. J Public Health Dent. 1996;56(3 Spec No):141-5; discussion 161-3. doi: 10.1111/j.1752-7325.1996.tb02424.x. PMID 8915959
- [Background] Oscarson N, Kallestal C, Fjelddahl A, Lindholm L. Cost-effectiveness of different caries preventive measures in a high-risk population of Swedish adolescents. Community Dent Oral Epidemiol. 2003 Jun;31(3):169-78. doi: 10.1034/j.1600-0528.2003.00033.x. PMID 12752542
- [Background] Ngo HC, Mount G, Mc Intyre J, Tuisuva J, Von Doussa RJ. Chemical exchange between glass-ionomer restorations and residual carious dentine in permanent molars: an in vivo study. J Dent. 2006 Sep;34(8):608-13. doi: 10.1016/j.jdent.2005.12.012. Epub 2006 Mar 15. PMID 16540227
- [Background] Miki S, Kitagawa H, Kitagawa R, Kiba W, Hayashi M, Imazato S. Antibacterial activity of resin composites containing surface pre-reacted glass-ionomer (S-PRG) filler. Dent Mater. 2016 Sep;32(9):1095-102. doi: 10.1016/j.dental.2016.06.018. Epub 2016 Jul 12. PMID 27417376
- [Background] Mickenautsch S, Yengopal V, Banerjee A. Atraumatic restorative treatment versus amalgam restoration longevity: a systematic review. Clin Oral Investig. 2010 Jun;14(3):233-40. doi: 10.1007/s00784-009-0335-8. Epub 2009 Aug 18. PMID 19688227
- [Background] Abanto J, Paiva SM, Sheiham A, Tsakos G, Mendes FM, Cordeschi T, Vidigal EA, Bonecker M. Changes in preschool children's OHRQoL after treatment of dental caries: responsiveness of the B-ECOHIS. Int J Paediatr Dent. 2016 Jul;26(4):259-65. doi: 10.1111/ipd.12192. Epub 2015 Sep 15. PMID 26370072
- [Background] Amaral MT, Guedes-Pinto AC, Chevitarese O. Effects of a glass-ionomer cement on the remineralization of occlusal caries--an in situ study. Braz Oral Res. 2006 Apr-Jun;20(2):91-6. doi: 10.1590/s1806-83242006000200001. PMID 16878198
- [Background] Anusavice KJ. Preservative dentistry: the standard of care for the 21st century. J Public Health Dent. 1995 Spring;55(2):67-8. doi: 10.1111/j.1752-7325.1995.tb02334.x. No abstract available. PMID 7643329
- [Background] Bonifacio CC, Hesse D, de Oliveira Rocha R, Bonecker M, Raggio DP, van Amerongen WE. Survival rate of approximal-ART restorations using a two-layer technique for glass ionomer insertion. Clin Oral Investig. 2013 Sep;17(7):1745-50. doi: 10.1007/s00784-012-0859-1. Epub 2012 Oct 11. PMID 23053709
- [Background] de Amorim RG, Leal SC, Frencken JE. Survival of atraumatic restorative treatment (ART) sealants and restorations: a meta-analysis. Clin Oral Investig. 2012 Apr;16(2):429-41. doi: 10.1007/s00784-011-0513-3. Epub 2011 Jan 28. PMID 21274581